CLINICAL TRIAL: NCT06720116
Title: Sustained Natural Apophysial Glide Versus Instrument Assisted Soft Tissue Mobilization in Patients With Chronic Mechanical Neck Pain
Acronym: MNP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Menna Allah Hesham Abd elfatah, principle investigator : menna allah hesham abd elfatah, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005464
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Mechanical Neck Pain
Keywords: Sustained Natural Apophysial Glide; instrument Assisted Soft Tissue Mobilization; Chronic Mechanical Neck Pain

STUDY DESIGN:
Intervention Model Description: mulligan and iASTM groups
Who Masked: Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- sustained natural apophysial glide (Experimental): patients will receive sustained natural apophysial glide( SNAGS ) in addition to conventional therapy in the form of ( Infrared, TENS , stretching exercices, isometric exercises) for chronic mechanical neck pain ,3 sessions per week for one month
  Interventions: Other: sustained natural apophysial glide; Other: conventional physical therapy
- instrument assisted soft tissue mobilization (Experimental): patients will receive instrument assisted soft tissue mobilization ( IASTM) technique in addition to conventional therapy in the form of ( Infrared, TENS , stretching exercices, isometric exercises) for chronic mechanical neck pain ,3 sessions per week for one month.
  Interventions: Other: instrument assisted soft tissue mobilization; Other: conventional physical therapy
- conventional therapy (Active Comparator): patients will receive conventional therapy in the form of ( Infrared, TENS , stretching exercices, isometric exercises) for chronic mechanical neck pain ,3 sessions per week for one month.
  Interventions: Other: conventional physical therapy

INTERVENTIONS:
Other: sustained natural apophysial glide — The patients will be in the sitting position and asked to move their head in the direction that particularly produces their symptoms. As the participant moves their head, the physiotherapist gently glides the painful vertebra anteriorly and sustains the glide through the movement.
  During the application of the glide, the participant should stay symptom free and is instructed to stop moving if any PAIN is produced. This movement was repeated for 10 times for 3 sets, The interval between the sets was 15 to 20 seconds.After mobilization subject had to perform same exercises as conventional group plus conventional physical therapy
  Arms: sustained natural apophysial glide
Other: instrument assisted soft tissue mobilization — The subject will be in comfortable sitting position leaning on a treatment table with the arm crossed to rest the head. After cleaning the skin of the subject and the blade with alcohol swabs, a lubricant (Vaseline) was applied, and a sweeping technique was used to apply a deep yet comfortable soft tissue mobilization on the upper trapezius from origin to insertion for approximately 3 min.
  First, M2T blade will be utilized to locate the precise locations of limitation in the affected muscles. Second, the M2T blade was put at 45 degree angle by using convex surface to apply gentle strokes along the muscle. Subjects were instructed that slight hyperemia on the skin is a normal feeling and should subside before the next session.
  Arms: instrument assisted soft tissue mobilization
Other: conventional physical therapy — the patients will receive conventional physical therapy in the form of Infrared, TENS , stretching exercices, isometric exercises

SUMMARY:
this study will be conducted to investigate the effect of sustained natural apophysial glide and Instrument assisted soft tissue mobilization on pain intensity, cervical range of motion and neck functional disability level in patients with chronic mechanical neck pain

DETAILED DESCRIPTION:
Neck pain is a common musculoskeletal disorder in the era of technology. The International Association for the Study of Pain (IASP) has defined neck pain as:"Pain perceived as arising from anywhere with in the region bounded superiorly by superior nuchal line, inferior by an unoriginally transverse line through the tip of first thoracic spinous process, and laterally by saggital plane tangential to the lateral border of neck. Mulligan pioneered specific manual approach called mobilization with movement (MWM).The advance of this approach was aimed for application on the spinal joints. He claimed that his technique could improve the spinal range of motion (ROM) and decrease pain through the correction of a positional fault occurring between the surfaces of the involved facet joints. The most commonly used Mulligan technique is called "sustained natural apophyseal glides" or SNAGs, this technique has introduced in 1999 by Mulligan and is performed by applying an accessory glide along the axis of the facet joint of the affected level while the patient is doing an active movement from weight-bearing position. The pressure applied by the therapist in a cephalad direction over the spinous process (centrally) or the transverse process (unilaterally) or to the articular pillar of the affected vertebra.The IASTM therapy is designed to promote the restart of connective tissues by resorbing extra fibroses, encouraging collagen secondary to fibroblast recruited healing. In turn this leads to scar tissues, adhesions, and fascial limitations being released and broken down. M2t blade is a multifunctional instrument invented by Adam Bro ger that is reasonable in price and has many planes that can be used in treatment. Its efficiency in improving patients symptoms was proven through many studies. sixty patients with mechanical neck pain will be assigned randomly into three equal group; group A will receive mulligan plus traditional, group B will receive IASTM plus traditional and group C will receive traditional only

ELIGIBILITY:
Inclusion Criteria:

* Sixety patients of chronic mechanical neck pain diagnosed and reffered from physicians will be participants in the study .
* Patients of both genders will be included.
* The age of the participants will beranged from 20 and 55 years
* The BMI ranged between 18.9 and 25 kg/m2
* All patients who suffered from neck pain more than 3 months.

Exclusion Criteria:

* Malignancy
* cervical and cranial surgery
* Recent fractures
* spinal tumors
* severe disc herniation
* uncontrolled hypertension
* Heart Disease ( arrhythmia, pacemaker).
* Pregnant and breast feeding women.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
neck disability | up to four weeks
  Assessment of neck disability will be performed by Arabic version of neck disability index .It is valid and reliable tool in the assessment of neck function. The NDI can be calculated as a raw score or as a percentage Each segment is graded on a scale of 0 to 5, with 0 representing "no discomfort" and 5 suggesting "the most excruciating pain imaginable." With a maximum score of 50 as following

SECONDARY OUTCOMES:
pain intensity | up to four weeks
  pain intensity will be measured by visual analogue scale. It is a 10-cm (100-mm) line; with 0 refer to no pain while 100mm refer to extreme pain. Patients were requested to place a mark along the line to express their level of pain. The reliability VAS is moderate to good in subjects with musculoskeletal conditions.
cervical range of motion | up to four weeks
  cervical range of motion device will be used to measure the neck ROM for flexion, extension, rotations, and lateral flexion using 3 separate inclinometers which are attached to a plastic frame and secured to the head by Velcro strap and nose bridge. The sagittal plane inclinometer measures flexion - extension, the frontal plane inclinometer measures right and left lateral flexion, and the horizontal plane inclinometer with a magnetic neck collar measures right and left rotation.